CLINICAL TRIAL: NCT01719263
Title: Sequential Segmental Treatment of Emphysema With Upper Lobe Predominance (STEP-UP) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptake Medical Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-1570
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Emphysema
Keywords: emphysema; InterVapor; treatments; pulmonary rehabilitation; lung volume reduction; endoscopic lung volume reduction
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment plus Optimal Medical Therapy (Experimental): Patients will be treated with the InterVapor System and Optimal Medical Therapy
  Interventions: Device: InterVapor® treatment plus Optimal Medical Therapy
- Optimal Medical Therapy (Active Comparator): Patients will be treated according to Optimal Medical Therapy
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Device: InterVapor® treatment plus Optimal Medical Therapy — Patients will be treated with the InterVapor System in 1 to 2 segments in the upper lobes of each lung (2 to 3 segments total). Patients will also receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema are published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO GOLD workshop summary).
  Other Names: InterVapor or BTVA
  Arms: Treatment plus Optimal Medical Therapy
Other: Optimal Medical Therapy — Patients will receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema are published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO GOLD workshop summary).
  Arms: Optimal Medical Therapy

SUMMARY:
This study is designed to demonstrate safety and efficacy in patients with severe upper lobe predominant emphysema. For validity of the study, the results will be compared to patients that receive optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Heterogeneous emphysema with upper lobe predominance in both lungs
* FEV1 between 20% and 45% predicted
* Residual volume (RV) > 150% predicted
* Post-rehabilitation 6-minute walk test > 140 meters

Exclusion Criteria:

* More than 3 COPD related hospitalizations requiring antibiotics in past 12 months
* FEV1 < 20% predicted
* DLCO < 20% predicted or immeasurable DLCO
* Body mass index (BMI) < 18kg/m2 or > 32 kg/m2
* History of any of the following:

  * Left ventricular ejection fraction (EF) ≤ 40%
  * Stroke
  * Myocardial infarction or acute coronary syndrome in previous year
  * Hospitalization due to left ventricular failure in previous 3 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1-second (FEV1) compared to active comparator | Year 1
Quality of Life (SGRQ) | Year 1

SECONDARY OUTCOMES:
Responder rate for FEV1 % difference from baseline | Year 1
Responder rate SGRQ pts difference from baseline | Year 1
Responder rate 6MWD meter difference from baseline | Year 1
Lobar Volume Reduction HRCT | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, MD, Principal Investigator — Heidelberg University; Gregory Snell, MD, Principal Investigator — The Alfred Hospital, Melbourne, Australia
Locations (17):
- Australia (4):
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Otto-Wagner-Spital, Vienna, Austria
- Germany (9):
  - Charite Universitätsmedizin Berlin Campus Mitte, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe Berlin, Berlin
  - Asklepios Fachkliniken Gauting München, Gauting
  - Klinik Schillerhohe, Gerlingen
  - Universitätsklinik Halle, Halle
  - Asklepios Klinik Harburg, Hamburg
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Klinikum Nürnberg, Nuremberg
- Mater Misericordiae University Hospital, Dublin, Ireland
- Auckland City Hospital, Auckland, New Zealand
- Royal Bromptom & Harefield NHS Foundation, London, United Kingdom

REFERENCES:
- [Derived] Herth FJ, Valipour A, Shah PL, Eberhardt R, Grah C, Egan J, Ficker JH, Wagner M, Witt C, Liebers U, Hopkins P, Gesierich W, Phillips M, Stanzel F, McNulty WH, Petermann C, Snell G, Gompelmann D. Segmental volume reduction using thermal vapour ablation in patients with severe emphysema: 6-month results of the multicentre, parallel-group, open-label, randomised controlled STEP-UP trial. Lancet Respir Med. 2016 Mar;4(3):185-93. doi: 10.1016/S2213-2600(16)00045-X. Epub 2016 Feb 16. PMID 26899390
- [Derived] Bandyopadhyay S, Henne E, Gupta A, Barry R, Snell G, Strange C, Herth FJ. Segmental approach to lung volume reduction therapy for emphysema patients. Respiration. 2015;89(1):76-81. doi: 10.1159/000369036. Epub 2014 Dec 6. PMID 25500669
- [Derived] Valipour A, Herth FJ, Eberhardt R, Shah PL, Gupta A, Barry R, Henne E, Bandyopadhyay S, Snell G. Design of the randomized, controlled sequential staged treatment of emphysema with upper lobe predominance (STEP-UP) study. BMC Pulm Med. 2014 Dec 3;14:190. doi: 10.1186/1471-2466-14-190. PMID 25467378